CLINICAL TRIAL: NCT04308252
Title: Comparison of Microbiome Composition and Biomarkers in Pharmaco Resistant and Pharmaco-Sensitive Epilepsy
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor no longer pursuing Epilepsy development.
Sponsor: Senda Biosciences (Industry)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E-NEU-EPY-02
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Epilepsy in Children; Pharmaco-Resistant Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collecting blood and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pharmaco-resistant epilepsy (PRE): Pharmaco resistant patients are defined by seizures despite adequate dosing of ≥2 anticonvulsant drugs.
- Pharmaco-sensitive epilepsy (PSE): Pharmaco-sensitive patients are defined by no seizures for 6 months.
- Sibling control: Sibling of the of the PRE study participants.

SUMMARY:
The purpose of this study is to determine stool microbiome composition and biomarkers that are differentially abundant and those that are associated with response to treatment (eg, anticonvulsant drugs).

DETAILED DESCRIPTION:
Recent research suggests that the intestinal microbiota plays a central role in human health, and may play a role in a variety of central nervous system disorders, including seizure susceptibility. The microbiota has been shown to be associated with changes in factors relevant to neurotransmission, including neurotransmitter signaling, synaptic protein expression, long-term potentiation, and myelination. In addition to the microbiota's potential role in general neurotransmission, research suggests that the gut microbiome may differ between patients with pharmaco resistant and pharmaco-sensitive epilepsies. In support of this idea, ketogenic diet has been used as an alternative treatment for those with pharmaco-resistant epilepsy and there are indications of possible direct interactions of anti-epileptic drugs (AEDs) with the intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Study participant and/or legal representative is willing and able to give informed consent/assent for participation in the study.
* Study participant and/or legal representative is willing and able to comply with all study requirements, in the opinion of the Investigator.
* Study participant is between the ages of 12 and 21, inclusive, at the Screening Visit.
* Study participant resides at home (alone or with family).
* Study participant has a confirmed diagnosis of epilepsy (epilepsy groups only; not applicable to sibling controls).
* Study participant has continued unprovoked seizures despite trials of ≥2 appropriate antiepileptic drugs at therapeutic doses (pharmaco resistant epilepsy group only; not applicable to pharmaco sensitive epilepsy group or sibling controls).

Exclusion Criteria:

* Study participant has monogenic epilepsy.
* Study participant has a neurodegenerative disease, mitochondrial disease, metabolic disease, active central nervous system disease, active autoimmune disease, or active inflammatory bowel disease.
* Study participant is on, or has been on within 30 days prior to the Screening Visit, a ketogenic diet, low glycemic index diet, or modified Atkins diet therapy.
* Study participant has had surgery within 3 months of the Screening Visit.
* Study participant is a resident in a group or hospital setting.
* Study participant requires the use of a g-tube or formula feeding.
* Study participant has had antibiotic therapy within 60 days prior to the Screening Visit.
* Study participant has participated in the study of an investigational product within 3 months prior to the Screening Visit (or within 5 half lives of the investigational product, whichever is longer) or is currently participating in a study of an investigational product.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 150 study participants are planned, including approximately 50 pharmaco-resistant study participants, approximately 50 pharmaco sensitive study participants, and approximately 50 sibling controls of the pharmaco-resistant study participants.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Pharmaco-sensitive (PSE) vs. pharmaco-resistant epilepsy (PRE) defined by no seizures for 6 months, and seizures despite adequate dosing of ≥2 anticonvulsant drugs, respectively | 24 months
  Bacterial species and metabolomic biomarkers that are associated with PRE/PSE are determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided